CLINICAL TRIAL: NCT01372384
Title: Phase II, Open-label Study of Erlotinib (Tarceva®) Treatment in Patients With Locally Advanced, Metastatic or Recurrent Non-small Cell Lung Cancer Who Present Activating Mutations in the Tyrosine Kinase Domain of the Epidermal Growth Factor Receptor
Brief Title: A Study of Tarceva (Erlotinib) in Patients With Locally Advanced, Metastatic or Recurrent Non-Small Cell Cancer Who Present Epidermal Growth Factor Receptor Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25423
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150 mg orally daily

SUMMARY:
This open-label study will assess the efficacy and safety of Tarceva (Erlotinib) in patients with locally advanced, metastatic or recurrent non-small cell lung cancer who have not received previous chemotherapy for their disease and who present epidermal growth factor receptor mutations. Patients will receive Tarceva 150 mg orally daily until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Locally advanced (Stage IIIB), metastatic (Stage IV) or recurrent non-small cell lung cancer with mutations in the tyrosine kinase domain of the epidermal growth factor receptor (EGFR)
* At least one measurable lesion according to RECIST criteria
* European Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate hematological, liver and renal function
* Patients with stable cerebral metastases who have received surgical or radiotherapy will be eligible

Exclusion Criteria:

* Previous chemotherapy or therapy against EGFR for metastatic disease (neoadjuvant or adjuvant therapy after radical surgery is allowed if finalized >/= 6 months before entering the study)
* History of another neoplasm except for carcinoma in situ of the cervix, adequately treated basal cell skin carcinoma, radically treated prostate carcinoma with good prognosis (Gleason </= 6), or another curatively treated neoplasm without evidence of disease in the last 5 years
* Symptomatic cerebral metastases
* Any significant ophthalmologic abnormality
* Use of coumarins
* Pregnant or breast-feeding women
* Pre-existing parenchymal lung disease such as pulmonary fibrosis, lymphangiosis and carcinomatosis (if this is the only presence of the disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Bulgaria (5):
  - Plovdiv
  - Sofia
  - Stara Zagora
  - Varna
  - Veliko Tarnovo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In all 145 participants were screened, of these 6 participants were randomized; major reason for screen failure was negative mutation status.
Groups:
- Erlotinib: Participants received recommended dose of Erlotinib (150 mg/day). No dose escalation of erlotinib was permitted. Participants were treated until disease progression, unacceptable toxicity, death or participant request for discontinuation.
Period: Overall Study
Arm/Group | Erlotinib
Started | 6
Completed | 3
Not Completed | 3
Not completed — Progression of disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (Tumour Assessments According to RECIST Criteria)
Description: Progression free survival is (PFS) defined as the time from the first dose of Erlotinib to the date of first occurrence of disease progression or death.
Time Frame: Until participants had disease progression, unacceptable toxicity or died; approximately 24 months.
Population: The Intent-to-treat (ITT population) included all patients with at least one valid post-baseline assessment.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Erlotinib
Number analyzed (Participants) | 6
Days | 223 [137 to 297]

2. Secondary Outcome: Objective Response Rate (Investigator Assessed)
Description: Objective response rate (ORR) was defined by RECIST criteria: Partial response (PR) was defined as ≥ 30% decrease in the sum of longest diameter of all target lesions, from the baseline sum. Complete response (CR) was defined as disappearance of all target and non-target lesions. For CR or PR, tumor measurements must be confirmed by 2nd assessments within 4 weeks. Progression of disease (PD) = 20% increase in the sum of longest diameter of all target lesions, from smallest sum of longest diameter of all target lesions recorded at or after baseline; or a new lesion; or progression of non-target lesions. Stable Disease (SD) = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on the study.
Time Frame: Visit 4, Visit 6, Visit 10 and Visit 22; (up to approximately 24 months)
Population: The ITT population included all patients with at least one valid post-baseline assessment. Only those participants available at the specified time points were analyzed (represented by n=X).
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Erlotinib
Number analyzed (Participants) | 6
Percentage
  Visit 4, SD, n=5 | 83.3 [35.87 to 99.58]
  Visit 4, PR, n=1 | 16.7 [0.42 to 64.13]
  Visit 6, SD, n=2 | 33.3 [4.32 to 77.73]
  Visit 6, PR, n=2 | 33.3 [4.32 to 77.73]
  Visit 6, PD, n=2 | 33.3 [4.32 to 77.73]
  Visit 10, PR, n=2 | 33.3 [4.32 to 77.73]
  Visit 10, PD, n=4 | 66.7 [22.27 to 95.68]
  Visit 22, PD, n=6 | 100 [0 to 100]
Statistical Analysis 1: Comparison: Erlotinib; Response assessment of Stable Disease Vs Partial Response at Visit 4 (Two proportions for Stable Disease Vs Partial Response of Erlotinib): The observed significance value of performed test for differences between two proportions for Stable Disease Vs Partial Response was analyzed; Test type: Superiority or Other; p = 0.045, Clopper-Pearson "exact" method
Statistical Analysis 2: Comparison: Erlotinib; Response assessment of Stable Disease Vs Partial Response at Visit 6 (Two proportions for Stable Disease Vs Partial Response of Erlotinib): The observed significance value of performed test for differences between two proportions for Stable Disease Vs Partial Response was analyzed; Test type: Superiority or Other; p = 1.000, Clopper-Pearson "exact" method
Statistical Analysis 3: Comparison: Erlotinib; Response assessment of Partial Response Vs Progression of disease at Visit 6 (Two proportions for of Partial Response Vs Progression of disease of Erlotinib): The observed significance value of performed test for differences between two proportions for of Partial Response Vs Progression of disease was analyzed; Test type: Superiority or Other; p = 1.000, Clopper-Pearson "exact" method
Statistical Analysis 4: Comparison: Erlotinib; Response assessment of Stable Disease Vs Progression of disease at Visit 6 (Two proportions for of Stable Disease Vs Progression of disease of Erlotinib): The observed significance value of performed test for differences between two proportions for of Stable Disease Vs Progression of disease was analyzed; Test type: Superiority or Other; p = 1.000, Clopper-Pearson "exact" method
Statistical Analysis 5: Comparison: Erlotinib; Response assessment of Partial Response Vs Progression of disease at Visit 10 (Two proportions for of Partial Response Vs Progression of disease of Erlotinib): The observed significance value of performed test for differences between two proportions for of Partial Response Vs Progression of disease was analyzed; Test type: Superiority or Other; p = 0.274, Clopper-Pearson "exact" method

3. Secondary Outcome: Safety: Incidence of Adverse Events
Description: An AE is any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. An SAE is any experience that suggests a significant hazard, contraindication, side effect, or precaution.
Time Frame: Until participants had disease progression, unacceptable toxicity, or died; approximately 24 months.
Population: All participants who received at least one dose of study medication and had a safety assessment performed post baseline were included in the safety population. Participants were analyzed according to the first dose received during the study.
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 6
participants
  Any AE | 6
  SAE | 1

4. Secondary Outcome: Overall Survival
Description: The overall survival (OS) is defined as the time from the first dose of Erlotinib to the date of death due to any cause.
Time Frame: Until participants had disease progression, unacceptable toxicity, or died; approximately 24 months.
Population: The ITT population included all patients with at least one valid post-baseline assessment.
Measure: Median (Full Range); unit: Days
Arm/Group | Erlotinib
Number analyzed (Participants) | 6
Days | 401 [160 to 670]

ADVERSE EVENTS:
Time Frame: Upto 24 months
Description: Serious adverse events and non-serious adverse events are reported in Safety Analysis Set, which consists of all participants who received at least one dose of study medication and had a safety assessment performed post baseline.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=6)
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=6)
Blood bilirubin increased (Investigations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Keratitis (Eye disorders) | 1
Orchitis (Reproductive system and breast disorders) | 1
Candidiasis (vulvovaginal) (Reproductive system and breast disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1
Parasternal pain (Musculoskeletal and connective tissue disorders) | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 2
Abnormal weight gain (Metabolism and nutrition disorders) | 1
Forunculosis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.